CLINICAL TRIAL: NCT07288853
Title: Mobile Application Push Notification in Improving Oral Hygiene Behaviour in Adolescent Orthodontic Patients: a Randomized Controlled Trial
Brief Title: Mobile Application Push Notification in Improving Oral Hygiene Behaviour in Adolescent Orthodontic Patients
Acronym: IMGS_EZGIGI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kumeran A/L Mohan (Other)
Collaborators: International Islamic University Malaysia (Other)
Responsible Party: Sponsor-Investigator, Kumeran A/L Mohan, Asst Prof Dr, International Islamic University Malaysia
Organization: International Islamic University Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IMGS25-003-0003
Record Dates: First submitted 2025-11-24; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Dental Plaque and Gingivitis; Oral Hygiene Reinforcement During Fixed Orthodontic Treatment
Keywords: push notification; oral hygiene reinforcement; fixed orthodontic treament; orthodontic plaque index (OPI); gingival index
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ezgigi with push notification (Experimental): Using mobile app EzGigi WITH DAILY PUSH NOTIFICATION to explain post bond up instructions and advice to watch daily videos posted on oral hygiene instructions and dietary advice
  Interventions: Behavioral: Ezgigi with push notification
- Ezgigi (Experimental): Using mobile app EzGigi to explain post bond up instructions and advice to watch daily videos posted on oral hygiene instructions and dietary advice
  Interventions: Behavioral: EzGigi
- conventional chairside post bond up instruction (No Intervention): Standard chairside post bond up instructions and advice on oral hygiene instructions and dietary advice

INTERVENTIONS:
Behavioral: Ezgigi with push notification — Using mobile app EzGigi WITH DAILY PUSH NOTIFICATION to explain post bond up instructions and advice to watch daily videos posted on oral hygiene instructions and dietary advice
  Arms: Ezgigi with push notification
Behavioral: EzGigi — Using mobile app EzGigi to explain post bond up instructions and advice to watch daily videos posted on oral hygiene instructions and dietary advice
  Arms: Ezgigi

SUMMARY:
This research looks at whether using a mobile phone app that sends push-notification reminders can help adolescent orthodontic patients keep their teeth and gums cleaner during treatment.

When teenagers wear braces, it's easy for food and plaque to get stuck around brackets and wires, which can lead to gingivitis and white spot lesions if oral hygiene isn't maintained. Traditional reminders from dentists often fade over time, so this study tests a more consistent, digital approach.

The app sends daily notifications reminding users to brush and care for their teeth. The study will compare three groups:

App with push-notification reminders,

App without reminders, and

Control group with normal instructions only.

Researchers will measure changes in plaque and gum health and use a questionnaire to see if the reminders also improve patients' knowledge, attitude, and practice (KAP) about oral hygiene.

In simple terms, the project tests if short smartphone reminders can make orthodontic patients more consistent, informed, and motivated in caring for their teeth.

DETAILED DESCRIPTION:
General objective:

To evaluate the effectiveness of push notification oral hygiene reminders on oral hygiene improvement and behavioural changes

Specific objectives:

To evaluate the oral hygiene improvement using push notification in a mobile phone application To assess the improvement in knowledge, attitude and practice (KAP) towards oral hygiene using push notification reminders in a mobile phone application

Study Design This is a 3-arm parallel-group randomized controlled trial (RCT) to evaluate the effectiveness of push notification-based oral hygiene reminders on oral hygiene improvement and behavioural changes among orthodontic patients with fixed appliances.

Trial setting The will be single centred study conducted in the Postgraduate Orthodontic Clinic, International Islamic University Malaysia, Kuantan Campus.

Ethical consideration Ethics approval will be acquired from the IIUM Research Ethics Committee (IREC) before study commencement. This study will also be in line with the CONSORT guidelines. Written informed consent will be obtained from each participant, ensuring full comprehension of study aims, procedures, risks, and benefits. Participants' data confidentiality will be maintained, adhering to the Declaration of Helsinki.

Eligibility criteria Inclusion criteria Exclusion criteria Aged 12-18 years Suitable for upper and lower arch fixed appliance treatment Good oral hygiene Able to understand Bahasa Malaysia and/or English Possess a personal or parental smartphone with app access Medically compromised or syndromic patients Need to skip bracket bonding On antibiotics Undergoing periodontal therapy Already using another dental reminder or behavior-change app Patients with cognitive or developmental limitations preventing app use

Intervention and comparator Arm 1: Access to the EzGiGi app, and daily behavioural and motivational push notification reminders Arm 2: Access to the EzGiGi app only Arm 3: No digital intervention Conduct of study Eligible patient will be identified through screening during initial pre-orthodontic assessment by the treating orthodontists or postgraduate orthodontic residents, during which relevant records such as a thorough intraoral assessment of dental and gingival health, intraoral and extraoral photographs, study models, and radiographs (dental panoramic radiographs and lateral cephalometric radiographs) are taken.

Upon selection, and obtaining informed consent, patient will be allocated to a randomly assigned treatment group. Fixed appliance treatment commences with upper and lower arch bond up using conventional metal brackets and round Nickel Titanium archwires. The patient will be required to complete a KAP questionnaire. Post operative instructions are then given, with the assigned mode of oral health knowledge reminder, according to their allocated group.

Patients' follow up visits are every 6 weeks. During these visits, Plaque Index and Gingival Index are also done at 6, 12, 18, 24 weeks. A follow-up KAP questionnaire on the patient's dental health knowledge is also done at 24 weeks. Once the study closes out, the fixed appliance treatment will be continued to completion.

Outcomes

Primary outcomes Orthodontic Plaque Index The Orthodontic Plaque index is used to assess the amount of dental plaque which accumulates around the bracket and bands of a fixed appliance. The index consists of scoring system as below.

Score 0: No plaque visible around bracket. Score 1: Plaque covering less than 1/3 of the bracket area. Score 2: Plaque covering between 1/3 and 2/3 of the bracket area. Score 3: Plaque covering more than 2/3 of the bracket area.

Patients will first be asked to chew on a disclosing tablet to identify the plaque clearly. An accumulated score is taken from 6 teeth (16, 11, 25, 36, 31, 45) and then averaged to conclude an overall plaque index value. If any of the teeth mentioned has been extracted, then the adjacent tooth will be used.

This step will be done during baseline, week 6, 12, 18 and 24.

Gingival Index The Gingival Index is a widely used measurement tool to assess gingival health of patients. Assessment is done based on colour, oedema and bleeding on probing. The index consists of the following scoring system.

Score 0: Normal gingiva (no inflammation pink firm). Score 1: Mild inflammation (slight change in color slight edema no bleeding on probing).

Score 2: Moderate inflammation (redness edema glazing bleeding on probing). Score 3: Severe inflammation (marked redness edema ulceration spontaneous bleeding).

The assessment will be done based on the visual assessment (to assess colour and oedema) and gingival probing using a periodontal probe (to assess spontaneous or delayed bleeding on probing) This step will be done during baseline, week 6, 12, 18 and 24.

Secondary outcomes Knowledge, Attitude and Practice questionnaire The KAP Questionnaire on Oral Hygiene and Interdental Cleaning is a validated, bilingual, self-administered questionnaire where questions will be marked (correct or incorrect). Finally, the accumulated percentage will be calculated. This questionnaire will be administered during baseline and at 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12-18 years
* Suitable for upper and lower arch fixed appliance treatment
* Good oral hygiene
* Able to understand Bahasa Malaysia and/or English
* Possess a personal or parental smartphone with app access

Exclusion Criteria:

* Medically compromised or syndromic patients
* Need to skip bracket bonding
* On antibiotics
* Undergoing periodontal therapy
* Already using another dental reminder or behavior-change app
* Patients with cognitive or developmental limitations preventing app use

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Gingival health | 6, 12, 18 and 24 weeks
  Assess Gingival Index using the scale below:
  0 Normal gingiva: pink, firm, no inflammation, no bleeding.
  1. Mild inflammation: slight color change, slight edema, no bleeding on probing.
  2. Moderate inflammation: redness, edema, glazing, bleeding on probing.
  3. Severe inflammation: marked redness, edema, ulceration, spontaneous bleeding.
  8 teeth (4 on each arch) will be assessed on all patients. The points are accumulated to assess the gingival condition.
Plaque amount | 6, 12, 18 and 24 weeks
  Orthodontic Plaque Index will be assessed using the following:
  0 No visible plaque.
  1. Thin film of plaque detected only by running a probe/explorer.
  2. Visible plaque covering less than one-third of the bracket area.
  3. Heavy plaque accumulation covering more than one-third of the area (thick, clearly visible deposits).
  patient's will be asked to chew on a disclosing tablet first, and 4 points will be assessed for each tooth:
  * Gingival area (margin)
  * Mesial area
  * Distal area
  * Occlusal/incisal area
    8 teeth will be assessed (4 each arch). The score is accumulated to assess plaque amount.

SECONDARY OUTCOMES:
Oral Hygiene and Interdental Cleaning | baseline and 24 weeks
  A validated questionnaire of "Knowledge, Attitude and Practice changes in oral hygiene and dietary advice" will be used, with each scored on a Likert scale (1-5). The total points will be calculated.

IPD SHARING:
Plan to Share IPD: No